CLINICAL TRIAL: NCT03344445
Title: Difference of Information Gain Between Video-base and Doctor Interview After Preanesthetic Visit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRB of NTUH Hsin-Chu Branch (Other)
Responsible Party: Sponsor-Investigator, IRB of NTUH Hsin-Chu Branch, Department of Anesthesia, National Taiwan University Hospital Hsin-Chu Branch
Organization: National Taiwan University Hospital Hsin-Chu Branch (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 102-019-E
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: simple compare of information gain between traditional visit and video-assisted visit
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional vist (No Intervention): Patients receive traditional anesthesiologist visit
- video-assisted (Experimental): Patients watch the video, then an anesthesiologist visit
  Interventions: Other: video-assisted pre anesthesia explain

INTERVENTIONS:
Other: video-assisted pre anesthesia explain — Anesthesiologist will visit all study patients, and only the experimental group will read the video.
  Arms: video-assisted

SUMMARY:
To investigate the differenec of patients' satisfaction and information gain betweem face-to-face interview and video introduction

DETAILED DESCRIPTION:
We made up a video which showed the type, the method, the risk, and the benefit of all anesthesia with words, pictures, and image. A study nurse will ask the will of patients. The patients enrolled in the study will be randomly divided into traditional group(control group) and study group(study group). The study group will watch the video at first, then our anesthesiologist visit the patient. The control group will receive traditional anesthesiologist visit. After doctors' visit, the patients have to complete a test and a questionnaire. The patients who don't participate in the study will have traditional visit and no test.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients were included who were scheduled to undergo elective surgery

Exclusion Criteria:

* Postoperative stay in the intensive care unit was expected or unexpected.,Repeated general anesthesia had been performed in the previous 6 months,ASA classification was more than or equal to III,There were pronounced cognitive and or speech barriers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
inform gain analysis | after every 100 effective data or 1 year, analyzed the data
  The score of test would represent the inform gain of patient
satification anaylsis | after every 100 effective data or 1 year, analyzed the data
  The score of questionnaire represent the ratification of patient

CONTACTS AND LOCATIONS:
Overall Officials: Li Kuei Chen, M.D., Study Chair — National Taiwan University Hospital Hsin-Chu Branch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang YL, Wang KJ, Chen WH, Chuang KC, Tseng CC, Liu CC. Improved satisfaction of preoperative patients after group video-teaching during interview at preanesthetic evaluation clinic: the experience of a medical center in Taiwan. Acta Anaesthesiol Taiwan. 2007 Sep;45(3):149-54. PMID 17972617
- [Result] Snyder-Ramos SA, Seintsch H, Bottiger BW, Motsch J, Martin E, Bauer M. Patient satisfaction and information gain after the preanesthetic visit: a comparison of face-to-face interview, brochure, and video. Anesth Analg. 2005 Jun;100(6):1753-1758. doi: 10.1213/01.ANE.0000153010.49776.E5. PMID 15920209